CLINICAL TRIAL: NCT03102671
Title: HeartHab: a Prospective Cross-over Trial Investigating the Effectiveness of an App Based Telerehabilitation Program on Exercise Capacity, Lifestyle and Risk Factors in Patients With Coronary Artery Disease
Brief Title: Effectiveness of the HeartHab Application on Exercise Capacity in Patients With Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, prof. dr. Paul Dendale, Principal Investigator, Hasselt University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HeartHab-002
Record Dates: First submitted 2017-03-26; First posted 2017-04-06 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AB sequence (Experimental): Usual care followed by use of HeartHab application: Treatment A comprises the usual care (i.e. one information session on the importance of medication adherence, risk factor control and healthy lifestyle), followed by telemonitoring during treatment B. The tele-intervention will consist of two months telerehabilitation and telecoaching concerning physical activity, healthy lifestyle and medication adherence.
  Interventions: Other: Usual care followed by the use of HeartHab application
- BA sequence (Experimental): Use of HeartHab application followed by usual care: patients will be followed by telemonitoring during treatment B. The tele-intervention will consist of two months telerehabilitation and telecoaching concerning physical activity, healthy lifestyle and medication adherence, followed by treatment A comprises the usual care (i.e. one information session on the importance of medication adherence, risk factor control and healthy lifestyle)
  Interventions: Other: Use of HeartHab application followed by usual care

INTERVENTIONS:
Other: Use of HeartHab application followed by usual care — use of a mobile, app based multidisciplinary telerehabilitation program (2 months) followed by usual care (two months)
  Arms: BA sequence
Other: Usual care followed by the use of HeartHab application — Usual care (2 months) followed by the use of HeartHab application (two months)
  Arms: AB sequence

SUMMARY:
The recurrence of major cardiac events after infarction is very high, in some populations up to 20% in the first year. Optimal secondary prevention as organized in cardiac rehabilitation centers is effective in reducing both morbidity and mortality. However, many studies have shown that the participation and adherence rate in CR-programs is low in most European countries. Therefore, novel ways of delivering secondary prevention using information technology and self-monitoring are being explored. Hence, this study will investigate the effectiveness of a mobile, patient tailored, app based multidisciplinary telerehabilitation program (HeartHab app) in improving exercise capacity, lifestyle and risk factors in patients with coronary artery disease in a post-rehabilitation setting.

DETAILED DESCRIPTION:
Study design and population This study is a prospective double-arm, non-pragmatic, cross-over, randomized controlled trial. Approximately 30 subjects will be selected retrospectively from the cardiology database of the Jessa Hospital Hasselt. Subjects who do not violate any of the predefined exclusion criteria and have provided informed consent will be randomly assigned in a 1:1 ratio to the treatment strategies (AB sequence or BA sequence).

After two months, each individual will be switched to the other treatment strategy.

Measurements At baseline, after two months (+14 days) and after four months (+14 days), a clinical assessment, medical history, current medication therapy, fasting blood sample, maximal cardiopulmonary exercise test, pulmonary function and three completed questionnaires (HeartQol, IPAQ and EQ-5D) will be collected of all patients. A fourth questionnaire will be completed by all the patients, focusing on the usability of the HeartHab-application.

Statistical analysis Data analysis will be performed using SPSS version 22 (SPSS Inc, Chicago, IL, USA) according to the intention-to-treat principle by assigned treatment group. Nonparametric alternatives will be used for parametric statistics in case assumptions for the latter are violated. The Shapiro-Wilk test will be used to assess normality. Paired t tests (parametric) or Wilcoxon signed rank tests (nonparametric) will be used for within-group analysis; independent t tests (parametric) or Mann-Whitney U tests (nonparametric) for between-group analysis. Chi-square tests will be used in case of categorical variables; Fisher's exact tests will be used when expected frequencies are small. The significance level for tests is 2-sided α=.05.

The cost-effectiveness evaluation will be conducted from a society and patient perspective, taking into account both intervention and health care resource costs. As the majority of patients will be retired, productivity losses due to illness-related absence from the workplace will not be taken into account.

Health care costs will be the aggregated costs of hospital admissions for cardiovascular reasons and also specialist visits and associated diagnostics. The cardiovascular rehospitalizations' related costs will be derived from invoices retrieved from the recruiting hospitals' financial departments. INAMI/RIZIV's nomenclature-based tariffs will define specialist visits and diagnostics denominations.

Quality adjusted life years (QALYs) will be used as a generic measure of effectiveness. Estimates of QALYs will be derived from the EQ-5D questionnaire. The EQ-5D scores will be converted to utility scores. The utility estimates will be converted to adjusted mean QALYs by calculating the area under the curve (AUC) utility estimates for all time intervals for each patient, weighted by the length of follow-up at that time interval. The change from baseline utility (adjusted differential incremental QALYs) will then be calculated, using the multiple regression model to control for baseline utility differences.

The incremental cost-effectiveness ratio (ICER) will be calculated (ICER¼(Cost intervention group - Cost control group)/(Effectiveness intervention group - Effectiveness control group)) to compare costs and outcomes (effectiveness) across both treatment groups. The incremental cost will be determined by the difference in total average cost per patient between the intervention group and control group. The incremental effectiveness will be estimated by the adjusted differential incremental QALYs.

ELIGIBILITY:
Inclusion Criteria:

* History of coronary artery disease with or without intervention (PCI/CABG/conservative)
* History of a cardiac rehabilitation (CR) program
* Clinically stable without inducible ischemia or high risk ventricular arrhythmia, confirmed by the last available maximal ergospirometry test
* Age ≥18 years
* Willing and physically able to follow an app based telerehabilitation program and other study procedures in a four months follow-up period
* Evidence of a personally signed and dated informed consent, indicating that the subject (or legally-recognised representative) has been informed of all pertinent aspects of the study
* Possession of and/or able to use an Android smartphone
* Dutch speaking and understanding

Exclusion Criteria:

* Recent PCI or CABG procedure, and still included in a CR program
* Orthopedic, neurologic or any other pathologic condition which makes the patient physically unable to follow an app based telerehabilitation program
* Planned interventional procedure or surgery in the next four months
* Pregnant females
* Present cardiovascular complaints
* Participation in other cardiac rehabilitation program trials, focusing on exercise outcome
* Any condition which in the opinion of the investigator would make it unsafe or unsuitable for the patient to participate in this study or a life expectancy of less than 4 months based on investigators judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Change in VO2peak | day1
  Exercise capacity is defined as the peak oxygen uptake, measured by CPET (cardiopulmonary exercise test)
Change in VO2peak | month 2 + 14 days
  Exercise capacity is defined as the peak oxygen uptake, measured by CPET (cardiopulmonary exercise test)
Change in VO2peak | month 4 + 14 days
  Exercise capacity is defined as the peak oxygen uptake, measured by CPET (cardiopulmonary exercise test)

SECONDARY OUTCOMES:
Risk factor profile: physiological parameter | day 1
  Blood pressure
Risk factor profile: physiological parameter | day 1
  Diabetes
Risk factor profile: physiological parameter | day 1
  Overweight
Risk factor profile: physiological parameter | day 1
  Smoking
Risk factor profile: physiological parameter | day 1
  Physical activity
Risk factor profile: physiological parameter | month 2 + 14 days
  Blood pressure
Risk factor profile: physiological parameter | month 2 + 14 days
  Diabetes
Risk factor profile: physiological parameter | month 2 + 14 days
  Overweight
Risk factor profile: physiological parameter | month 2 + 14 days
  Smoking
Risk factor profile: physiological parameter | month 2 + 14 days
  Physical activity
Risk factor profile: physiological parameter | month 4 + 14 days
  Blood pressure
Risk factor profile: physiological parameter | month 4 + 14 days
  Diabetes
Risk factor profile: physiological parameter | month 4 + 14 days
  Overweight
Risk factor profile: physiological parameter | month 4 + 14 days
  Smoking
Risk factor profile: physiological parameter | month 4 + 14 days
  Physical activity
Generic health status: questionnaire | day 1
  EQ5D
Exercise capacity: questionnaire | day 1
  IPAQ
Quality of life: questionnaire | day 1
  Heart QoL
Generic health status: questionnaire | month 2 + 14 days
  EQ5D
Exercise capacity: questionnaire | month 2 + 14 days
  IPAQ
Quality of life: questionnaire | month 2 + 14 days
  Heart QoL
Generic health status: questionnaire | month 4 + 14 days
  EQ5D
Exercise capacity: questionnaire | month 4 + 14 days
  IPAQ
Quality of life: questionnaire | month 4 + 14 days
  Heart QoL
Cardiovascular events: clinical assessment | day 1
  Collection of adverse events during follow up visit
Cardiovascular events: clinical assessment | month 2 + 14 days
  Collection of adverse events during follow up visit
Cardiovascular events: clinical assessment | month 4 + 14 days
  Collection of adverse events during follow up visit

CONTACTS AND LOCATIONS:
Overall Officials: Paul Dendale, prof. dr., Principal Investigator — Hasselt University
Locations (1):
- Jessa Hospital, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sankaran S, Dendale P, Coninx K. Evaluating the Impact of the HeartHab App on Motivation, Physical Activity, Quality of Life, and Risk Factors of Coronary Artery Disease Patients: Multidisciplinary Crossover Study. JMIR Mhealth Uhealth. 2019 Apr 4;7(4):e10874. doi: 10.2196/10874. PMID 30946021